

## **Non-interventional Study Protocol**

| Document Number: | c19925296-03 |
|---|---|
| BI Study Number: | 1245.149 |
| BI Investigational Product(s): | Jardiance® (Empagliflozin) |
| Title: | Post-authorization safety study in patients with type 2 diabetes mellitus to assess the incidence of ketoacidosis, severe complications of urinary tract infection, volume depletion, and dehydration among patients treated with Empagliflozin or DPP-4 inhibitors in Saudi Arabia |
| Brief lay title | Post-authorization safety study in type 2 diabetic patients in Saudi Arabia treated with Empagliflozin to assess the incidence of ketoacidosis, severe complications of urinary tract infection, volume depletion, and dehydration |
| Protocol version identifier: | 3.0 |
| Date of last version of protocol: | 03 May 2018 |
| PASS: | Yes |
| EU PAS register number: | EUPAS20025 |
| Active substance: | Jardiance® (Empagliflozin 10mg & 25 mg) |
| Medicinal product: | Jardiance® film-coated tablets 10mg, 25mg |
| Product reference: | rence: Empagliflozin 10 mg: 103-68-16 |
| | Empagliflozin 25 mg: 104-68-16 |
| Procedure number: | SFDA application no. 17062102 on SCTR |
| Marketing authorisation holder(s): | Boehringer Ingelheim Saudi Arabia |
| Joint PASS: | No |
| Research question and objectives: | NIS with new data collection, with the following aims: Primary outcomes To estimate the incidence of |
| | To estimate the incidence of: - Ketoacidosis |
| | - Severe urinary tract infections |

| | Proprietary confidential information ternational GmbH or one or more of its affiliated companies. All rights reserved. part - be passed on, reproduced, published or otherwise used without prior written permission |
|---|---|
| | Page 1 of 42 |
| Date: | 23 Sep 2019 |
| Signature of EU-<br>QPPV: | The signature of the EU-QPPV is provided electronically |
| EU-QPPV: | |
| MAH contact person: | |
| Marketing authorisation holder: | Boehringer Ingelheim |
| Author: | |
| Country of study: | Multi-Centre study conducted in Saudi Arabia |
| | following definition of exposure: the Ramadan period |
| | Secondary outcomes To estimate the risk of each primary outcome with respect to the |
| | in type 2 diabetes mellitus (T2DM) patients exposed to Jardia (Empagliflozin) compared with the incidence in T2DM patier exposed to Dipeptidyl peptidase-4 (DPP-4) inhibitors |
| | - Dehydration |
| | - Volume depletion |

## 1. TABLE OF CONTENTS

| TITL | E PAG | E | 1 |
|------|---------|----------------------------------|----|
| 1. | TABLI | E OF CONTENTS | 3 |
| 2. | LIST C | F ABBREVIATIONS | 5 |
| 3. | RESPO | NSIBLE PARTIES | 7 |
| 4. | ABSTE | RACT | 8 |
| 5. | AMEN | DMENTS AND UPDATES | 13 |
| 6. | MILES | TONES | 14 |
| 7. | RATIC | NALE AND BACKGROUND | 15 |
| 8. | RESEA | RCH QUESTION AND OBJECTIVES | 16 |
| 8.1 | PRI | MARY OBJECTIVE | 16 |
| 8.2 | SEC | ONDARY OBJECTIVE | 16 |
| 9. | RESEA | RCH METHODS | 17 |
| 9.1 | STU | DY DESIGN | 18 |
| 9.2 | SET | TING | 18 |
| 9 | .2.1 | Study sites | 18 |
| 9 | .2.2 | Study population | 18 |
| | 9.2.2.1 | , | |
| | 9.2.2.2 | Visit 2; 16±2 weeks from Visit 1 | 20 |
| | 9.2.2.3 | Visit 3; 32±2 weeks from Visit 1 | 21 |
| | 9.2.2.4 | Visit 4; 52 weeks End of study | 21 |
| | 9.2.2.5 | 1 1 | |
| 9 | .2.3 | Study discontinuation | 22 |
| 9.3 | VAI | RIABLES | |
| 9 | .3.1 | Safety | 22 |
| | 9.3.1.1 | 3 | |
| | .3.2 | Exposures | |
| | .3.3 | Outcomes | |
| | .3.4 | Covariates | |
| 9.4 | | FA SOURCES | |
| 9.5 | | IDY SIZE | |
| 9.6 | DAT | ΓA MANAGEMENT | 27 |

| 9.7 | DA | TA ANALYSIS27 |
|------|--------|--------------------------------------------------------------|
| 9. | 7.1 | Propensity score modelling |
| 9. | 7.2 | Main analysis using stratification |
| 9.8 | _ | ALITY CONTROL |
| 9.9 | LIM | IITATIONS OF THE RESEARCH METHODS |
| 9.10 | OTI | HER ASPECTS |
| 9. | 10.1 | Data quality assurance |
| 9. | 10.2 | Study records |
| | 9.10.2 | .1 Source documents |
| | 9.10.2 | .2 Direct access to source data and documents |
| 10. | PROTI | ECTION OF HUMAN SUBJECTS |
| 10.1 | | JDY APPROVAL, PATIENT INFORMATION, AND INFORMED NSENT |
| 10.2 | STA | ATEMENT OF CONFIDENTIALITY |
| | | AGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE TIONS |
| 11.1 | DEI | FINITION OF ADVERSE EVENTS |
| 11.2 | | VERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND PORTING |
| 11.3 | REI | PORTING TO HEALTH AUTHORITIES |
| 12. | | S FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS |
| | | RENCES41 |
| 13.1 | PUI | BLISHED REFERENCES |

#### 2. LIST OF ABBREVIATIONS

ACR Albumin Creatinine Ratio

ADR Adverse Drug Reaction

AE Adverse Event

AESI Adverse Event of Special Interest

BI Boehringer Ingelheim

BP Blood Pressure

CA Competent Authority
CML Local Clinical Monitor

CRA Clinical Research Associate

CRO Contract Research Organization

CTP Clinical Trial Protocol
CTR Clinical Trial Report
DKA Diabetic ketoacidosis
DMP Data Management Plan
DPP-4 Dipeptidyl-peptidase 4

E-CRF Electronic Case Report Form

EDC Electronic Data Capture

eGFR Estimated Glomerular Filtration Rate

EU European Union

EU PAS European Union electronic register of post-authorization studies

EU-QPPV European Union-Qualified Person for Pharmacovigilance

FPG Fasting Plasma Glucose
GCP Good Clinical Practice
GLD Glucose lowering drug
GLUT Glucose Transporter

GPP Good Pharmacy Practice
HbA1c Glycated Hemoglobin

HDL-C High Density Lipoprotein Cholesterol

IC50 Inhibitory Concentration

ICH International Conference on Harmonisation

IEC Independent Ethics Committee

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

IRB Institutional Review Board

ISF Investigator Site File

LDL-C Low Density Lipoprotein Cholesterol

LPVM Local PV Manager

MAH Marketing Authorisation Holder Activities

MedDRA Medical Dictionary for Drug Regulatory Activities

MFDS The Ministry of Food and Drug Safety

SFDA Saudi Food & Drug Authority

#### 3. RESPONSIBLE PARTIES

Boehringer Ingelheim (BI) has appointed a Trial Clinical Monitor (TCM), responsible for coordinating all required activities, in order to

- Manage the study in accordance with applicable regulations and internal standard operating procedures (SOPs).
- direct the study team in the preparation, conduct, and reporting of the trial,
- order the materials as needed for the study,
- Ensure appropriate training and information of Local Clinical Monitors (CMLs), Clinical Research Associate (CRAs), and Investigators of Saudi Arabia.

The organization of the study will be done by a Contract Research Organization (with which the responsibilities and tasks will have been agreed and a written contract filed before initiation of the study. A CML will be appointed responsible for coordinating the activities required in order to manage the study in accordance with applicable regulations and internal SOPs in the countries covered by the respective BI OPU. On-site monitoring will be performed by a CRO appointed by BI.

An Investigator Site File (ISF) containing all relevant study related documentation will be maintained according to local regulations and BI and/or CRO SOPs at each study site. A copy of the ISF documents will also be kept as an electronic Trial Master File (TMF) at BI according to BI and/or CRO SOPs. Documents related to participating physician and other important participants, especially their curricula vitae, will be filed in the TMF.

## 4. ABSTRACT

| Name of company: | | | |
|---|---|---|---|
| Name of finished m<br>product:<br>Jardiance® | edicinal | | |
| Name of active ingr<br>Empagliflozin | edient: | | |
| Protocol date:<br>16 Oct 2017 | Study<br>number:<br>1245.149 | Version/Revision: 3.0 | Version/Revision date: 23 Sep 2019 |
| Title of study: | to assess the incitract infection, v | on safety study in patients wit idence of ketoacidosis, severe rolume depletion, and dehydra pagliflozin or DPP-4 inhibitor | complications of urinary ation among patients |
| Rationale and background: | According to the local regulations, for some safety concerns, additional pharmacovigilance activities, for instance post-authorization safety studies which are initiated, managed or financed by marketing authorization holders, voluntarily, or pursuant to obligations can be imposed by SFDA. SFDA has requested a non-interventional study (NIS) to provide supplementary data to monitor the safety of Jardiance® (Empagliflozin) in a real-life situation including the Ramadan period. | | |
| Research question and objectives: | Non-interventional study with new data collection, with the following aims: Primary outcomes To estimate the incidence of: - Ketoacidosis - Severe urinary tract infections - Volume depletion - Dehydration in type 2 diabetes mellitus (T2DM) patients initiating Jardiance® (Empagliflozin) compared with the incidence in T2DM patients initiating Dipeptidyl peptidase-4 (DPP-4) inhibitors Secondary outcomes To estimate the risk of each primary outcome with respect to the following definition of exposure: the Ramadan period Primary and secondary outcomes will be followed up for 1 year from Index date | | |

| Name of company: | | | |
|---|---|---|---|
| Name of finished mo<br>product:<br>Jardiance® | edicinal | | |
| Name of active ingredient:<br>Empagliflozin | | | |
| Protocol date:<br>16 Oct 2017 | Study<br>number:<br>1245.149 | Version/Revision: 3.0 | Version/Revision date: 23 Sep 2019 |
| Study design: | This will be non-interventional study with new data collection. The study will use a "new users" design and compare new users of Jardiance® (Empagliflozin) to new users of DPP-4 inhibitors. The index date will be defined as the date on which each identified new user receives the index prescription for Jardiance® (Empagliflozin) or a DPP-4 inhibitor. Number of recruited patients will be comparable in each group within a given timeframe (i.e. each site will ensure to recruit similar number of patients for each group according to assigned blocks of enrolment) Propensity scores based on information prior to the index date will be used to account for potential confounding. Patients will be follow-up for 12 months after index date. | | |
| Population: | Patients diagnosed with T2DM in Saudi Arabia The study population will include patients aged at least 18 years and diagnosed with T2DM in Saudi Arabia and who will initiate Jardiance® (Empagliflozin) treatment during the study period and who have not used other SGLT2 inhibitors during the previous 12 months. Patients switching to or adding Jardiance® (Empagliflozin) to other antidiabetic medications will be compared to patients switching to or adding comparator treatment on same background therapy. This modification of a "new-user" design is an appropriate method for studying second-line therapies in chronic conditions. The comparator groups will include new users of DPP-4 inhibitors. The same inclusion and exclusion criteria will be applied. Patients with a confirmed diagnosis of type 1 diabetes before or after the index date will not be included in the study. Patients prescribed fixed-dose combinations of SGLT2 inhibitors with DPP-4 inhibitors will be excluded. | | |

| Name of company: | | | |
|---|---|---|---|
| Name of finished n<br>product:<br>Jardiance® | nedicinal | | |
| Name of active ing<br>Empagliflozin | redient: | | |
| Protocol date:<br>16 Oct 2017 | Study<br>number:<br>1245.149 | Version/Revision: 3.0 | Version/Revision<br>date: 23 Sep 2019 |
| Variables: | Covariates: Variables potentially associated with outcomes of interest—such as Sociodemographic variables including age, sex, concomitant medications; will be identified for all cohort members prior to and including the index date. Severity of T2D will be assessed by HbA1c values concomitant diagnoses and duration since the first diagnosis, when available. These and other variables that can differ by exposure group will be considered for inclusion as predictors in the logistic regression models used to generate the propensity scores. Propensity scores will be used in the analysis to quantify the probability of receiving Jardiance® (Empagliflozin) at the index date for new users of both Jardiance® (Empagliflozin) and DPP-4 inhibitors. At the index date, cohort members will also be classified by indicator variables on the calendar time of cohort entry (by quarter) whether the index treatment (Empagliflozin or DPP-4 inhibitor) was added to existing medication (adding on), or if the index treatment was initiated as a replacement for another GLD (switching from the existing GLD to Jardiance® (Empagliflozin) or DPP-4 inhibitor, and whether this treatment was received as monotherapy or as dual or triple therapy. A variable indicating whether or not patients were receiving insulin at the index date will also be created. | | |
| Data sources: | The investigator will be asked to successively write in the case report forms (e-CRFs) from the subject who was initially administered the drug following the study start date to the requested number of subjects without omission. Data on the period preceding the index date will be collected at the time of the first survey. Prior to initiation of the study, written contract shall be concluded, and this contract shall be concluded with the head of the site or the investigator with his/her consent. Non-Interventional study with new data collection | | |
| Study size: | Based on the requirements of SFDA, the sample size will be 1500 patients overall, 750 patients in each group DPP4i and Empagliflozin. The recruitment process will be adjusted in each site accordingly. | | |

| Name of company: | | | |
|---|---|---|---|
| Name of finished m<br>product:<br>Jardiance® | nedicinal | | |
| Name of active ingr<br>Empagliflozin | redient: | | |
| Protocol date:<br>16 Oct 2017 | Study<br>number:<br>1245.149 | Version/Revision: 3.0 | Version/Revision<br>date: 23 Sep 2019 |
| Data analysis: | analysis will be corresponds to corresponds to contruction of the assessment data analysis wing the construction of the ketoacidosis dehydration con Additional sensitive robustness of alta and reduction of the following endergond the contruction of the following endergond the control of the following endergond the fo | ent of the primary and secondar II be conducted in two stages: of the propensity score (PS) by regaliflozin) vs. DPP-4 inhibitor the effect of exposure to Jardian and a severe urinary tract infections, appared to those exposed to DPP it intitity analyses will be performed ternative definitions of outcome of bias due to matching. Stimates and comparison will be usted incidence rates of each of pagliflozin) new users and amore rates will be reported as point of ears) and 95% confidence interves, after adjusting (via stratified pensity score deciles and calendar were versus DPP-4 inhibitors for each of the outcomes will be rest. Adjusted incidence rates are eighting the incidence or IRR of core decile and calendar year) by pagliflozin) person-time within analysis will further stratify the eindex date is stivity analyses will be performed. | l' (AT) approach. This ntinue use of the index ny other of the index ny other of the index ny other of the index ny other of the index ny objectives, the main modelling the exposure see (Empagliflozin) on ny volume depletion and ny volume depletion ny volume depletion ny volume depletion and ny volume depletion ny volume depletion and ny volume depletion and ny volume depletion and ny volume depletion ny volume depletion ny volume depletion ny volume depletion and ny volume depletion ny volume depletion and ny volume depletion |

| Name of company Name of finished product: Jardiance® | | | |
|---|---|---|---|
| Name of active in<br>Empagliflozin | gredient: | | |
| Protocol date:<br>16 Oct 2017 | Study<br>number:<br>1245.149 | Version/Revision: 3.0 | Version/Revision<br>date: 23 Sep 2019 |
| Milestones: | data through 12 | Data collection will start in Q3 2018; The Final report will be produced using data through 12 months from the start of use of Empagliflozin or DPP4I index date (currently planned study period data collection from Q3 2018 – Q4 2020). | |

## 5. AMENDMENTS AND UPDATES

| Number | Date | Section of study protocol | Amendment or update | Reason |
|---|---|---|---|---|
| 2.0 | 03 May 2018 | Milestones | Amendment | Shifting of study milestones due to delay of study initiation |
| 3.0 | 23 Sep 2019 | Milestones | Amendment | Extension of recruitment period |

## 6. MILESTONES

| Milestone | Planned Date |
|---|---|
| IRB/IEC approval | Q2 2018 – Q3 2018 |
| Start of data collection (trial data) FPI | Q3 2018 |
| Recruitment Period (LPI) | Q4 2019 |
| Ramadan Month 2019 | May 5th, $2019$ – June 4th, $2019 \pm 1-2$ days |
| Ramadan Month 2020 | April 23 <sup>rd</sup> , 2020 – May 23 <sup>rd</sup> , 2020 ±1-2 days |
| Interim Progress Report to<br>SFDA (as per the Saudi FDA<br>templates) | Q4 2018, Q2 2019, Q4 2019, Q2 2020, Q4 2020 |
| End of data collection ( LPV) | Q4 2020 |
| Final report of study results:<br>CSR preparation | Q2 2021 |

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 7. RATIONALE AND BACKGROUND

Around 415 million patients are affected by DM worldwide. DM is considered an epidemic in many countries of the world, and the number of people affected is expected to double over the next decade. [R16-4703] DM is a major leading cause of many complications and diseases such as heart diseases and several types of infections. T2DM is more common than type 1, comprising 90-95% of all DM cases. [R17-3422] Over 5 million people died from DM in 2015 worldwide. In the Middle East and North Africa, around 36 million patients were affected by DM in 2015, a number expected to rise to 72 million patients by 2040. Saudi Arabia has one of the highest prevalence of DM in the world with over 20% of the population affected. [R16-4703]

Empagliflozin is a selective sodium/glucose co-transporter 2 (SGLT2) inhibitors one of the most recent classes of drugs used to treat T2DM. SGLT2 inhibitors promote the renal excretion of glucose and help lower elevated blood glucose levels in patients with T2DM. [P14-06594] In Saudi Arabia, It is indicated for treatment of T2DM as monotherapy or addon combination therapy. It is used as monotherapy when exercise and diet control alone do not provide glycaemic control in patients for whom use of metformin is considered inappropriate because of intolerance. It is also used in combination with other glucose lowering agents—including insulin—when they do not provide adequate glycaemic control. [R17-3413] Several clinical trials showed the efficacy of Empagliflozin in reducing the blood glucose level. Furthermore, Empagliflozin is a unique drug among all hypoglycaemic agents because it has shown a reduction in major cardiovascular events, which has not been the case with other oral hypoglycaemic agents. Empagliflozin, as other SGLT2 inhibitors, is associated with some adverse reactions such as urinary tract infections and genital infections, especially in females. In addition, rare cases of diabetic ketoacidosis (DKA) have been reported. [P15-03461], [P13-09179], [P15-05613] In parallel to the launch of SGLT2 inhibitors in Saudi Arabia, the Saudi Food and Drug Authority (SFDA) has requested a noninterventional study to further monitor the safety of Empagliflozin in the country, including during the Ramadan period.

The objectives of this study are to assess the risk of ketoacidosis, severe urinary tract infections, volume depletion, and dehydration associated in patients with T2DM initiating Empagliflozin compared to patient initiating a dipeptidyl peptidase-4 (DPP-4) inhibitors over a 12-month period of follow-up, including the month of Ramadan.

#### 8. RESEARCH QUESTION AND OBJECTIVES

#### 8.1 PRIMARY OBJECTIVE

Non-interventional study with new data collection, with the following aims:

#### Primary outcomes

To estimate the incidence of:

- Ketoacidosis
- Severe urinary tract infections
- Volume depletion
- Dehydration

in T2DM patients initiating Empagliflozin compared with the incidence in T2DM patients initiating Dipeptidyl peptidase-4 (DPP-4) inhibitors.

#### 8.2 SECONDARY OBJECTIVE

To estimate the risk of each primary outcome with respect to the following definition of exposure:

- The Ramadan period

(1st day of Ramadan to 29th day of Ramadan based on the Islamic Hijri calendar)



Figure 1: Ramadan period during study follow-up time

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9. **RESEARCH METHODS**

This is a non-interventional study with new data collection.

This study will cover the period between Q3 2018 and Q4 2020. The main goals of this study are to examine the risk of ketoacidosis, severe urinary tract infections, volume depletion, and dehydration associated with the use of Empagliflozin compared to the use of DPP-4 inhibitors in T2DM patients. The study will use an "incident users" design and compare new users of Empagliflozin with new users of DPP-4 inhibitors. The index date will be defined as the date on which each identified new user receives the index prescription for Empagliflozin or DPP-4 inhibitors. The definition of drug exposure for Empagliflozin will be any patient using at least one prescription of Empagliflozin tablets (10 or 25 mg) or fixed-dose combinations with metformin. The comparator group will be comprised of patients with at least one prescription of a DDP-4 inhibitor: sitagliptin, saxagliptin, linagliptin, vildagliptin, alogliptin (and fixeddose combinations of these drugs with metformin). Each member of the population exposed to Empagliflozin must have at least one prescription for Empagliflozin, with or without other Glucose-lowering Drugs (GLDs,) and no prior prescriptions of a DPP-4 inhibitor or Empagliflozin during the available pre-index period. Each member of the population exposed to a DPP-4 inhibitor must have at least one prescription for a DPP-4 inhibitor, with or without other GLDs, and no prior prescriptions of a DPP-4 inhibitor or Empagliflozin during the available pre-index period.

Follow-up will start the day after the index date and will continue until any of the following conditions are met: date of death or after 12 months of follow-up, or the date during follow-up that specific exclusion criteria are met, the date of the last continuous treatment of the index drug (Empagliflozin or DPP-4 inhibitor) plus a defined grace period (30 days after the end of the last prescription's days' supply in main analyses), or the date in which a new treatment episode starts with any of the other index drugs. Patients who discontinue an index drug and then subsequently initiate another index drug will not be allowed to re-enter the study. Patients will be followed-up for 12 months.

This study will be carried out in the manner of successive surveys that the investigator will be asked to successively write in the case report forms (e-CRFs) from each subject who was initially administered the drug following the study start date until the requested number of subjects is reached. Number of recruited patients will be comparable in each group within a given timeframe (i.e. each site will ensure to recruit similar number of patients for each group according to assigned blocks of enrolment).

Prior to initiation of the study, a written contract shall be concluded, and this contract shall be executed among BI OPU, CRO with the head of the site or the investigator with his/her consent.

Patients will be managed according to the local practice guidelines. The choice of treatment will be solely at the discretion of the participating physician. Empagliflozin and the comparator DPP-4 inhibitor will be administered according to the approved labels in Saudi Arabia. [R17-3427] Hence there are no additional risks to patients by participating in this PASS.

#### 9.1 STUDY DESIGN

This is a non-interventional study with new data collection from T2DM patients in Saudi Arabia. The study will use a "new users" design and compare new users of Empagliflozin to new users of DPP-4 inhibitors in T2DM patients. We have chosen DDP-4 inhibitors because they are considered one of the new groups of hypoglycaemic agents, and they are one of the options to treat patients with T2DM as they have similar indications to Empagliflozin.

Number of recruited patients will be comparable in each group within a given timeframe (i.e. each site will ensure to recruit similar number of patients for each group according to assigned blocks of enrolment).

The index date will be defined as the date on which each identified new user receives the index prescription for Empagliflozin or DPP-4 inhibitors. The patients will be followed up for 12 months after the index date.

The incident-user design avoids comparing a population predominantly composed of first-time users of a newly marketed drug such as Empagliflozin with a population of prevalent users of an older drug who may have stayed on the comparator treatment for a longer time and be less susceptible to the events of interest.

Empagliflozin and the comparator DPP-4 inhibitor will be prescribed according to the local label and at the discretion of the treating physician. [R17-3427] Since this is a non-interventional study, the drug will not be supplied by the sponsor. Furthermore, the sponsor will not cover the expenses related to other medications taken by the patient, interventions, procedures, or diagnostic test.

#### 9.2 SETTING

#### 9.2.1 Study sites

A total of 1500 patients will be enrolled at approximately 25 sites in Saudi Arabia. The treating physicians will mainly be general practitioners (GPs) and/or specialists including endocrinologist, diabetologist & internists. Number of recruited patients will be comparable in each group within a given timeframe (i.e. each site will ensure to recruit similar number of patients for each group according to assigned blocks of enrolment).

#### 9.2.2 Study population

Main diagnosis for study entry

Patients diagnosed with T2DM will be included.

#### Inclusion criteria:

- Patients who have signed Informed consent form.
- The patients will be at least 18 years old at index date, diagnosed with T2DM in Saudi Arabia, and who will initiate Empagliflozin or DPP4 inhibitors treatment according to the local label and at the discretion of the treating physician during the study period, who have not used other SGLT2 or DPP4 inhibitors during the previous 12 months.

#### Exclusion criteria:

- Known hypersensitivity to Empagliflozin, the comparator DPP-4 inhibitors or any of their excipients
- Patients for whom Empagliflozin or the comparator DPP-4 inhibitor is contraindicated according SFDA approved label
- Patients prescribed fixed-dose combinations of SGLT2 inhibitors with DPP-4 inhibitors will be excluded.
- The same inclusion and exclusion criteria will be applied to the comparator group, which will include new users of DPP-4 inhibitors.



<sup>\*</sup> From Visit 1

Figure 2: Study Visits

#### **Baseline Visit**

#### 9.2.2.1 Visit 1; Baseline Visit

Upon patient enrolment, the following available data will be recorded on the patient's e-CRF.

- Visit date
- Diagnosis: date of the diagnosis of T2DM, Family history of T2DM
- Inclusion / Exclusion criteria

- Informed consent form: Date of Informed consent
- Demographic data: Age, gender,
- Diabetes mellitus related complication (Retinopathy, Neuropathy, Nephropathy)
- Medical history: Hypertension, Dyslipidaemia, Coronary artery disease, Stroke, Liver disease, Renal failure, Renal Transplant, Renal Stones Nephropathy, Prostate Diseases, Pancreatitis, Diabetic ketoacidosis, Surgery, Infections (other than UTIs) and heart diseases, other (history of concomitant disease within 6 months). In addition, genital defects, urinary tract anatomical defects, when available.
- Baseline lab variables when available Complete Blood Count (CBC), Oral Glucose Tolerance Test (OGTT), ketones level, amylase, lipase, arterial blood gas, pH, bicarbonate, lipid profile tests, Blood Urea Nitrogen (BUN), liver tests, International Normalized Ratio (INR) for prothrombin time and platelets
- Physical examination: body mass index (BMI), blood pressure, pulse rate, weight
- Baseline HbA1C, blood glucose level (if available)
- Renal Function: record Serum creatinine, eGFR, urine ACR if results are available (collected within the latest 2month period) (if available)
- Concomitant anti-hyperglycemic agent: record any anti-hyperglycemic agents have been taken prior to the baseline visit (within 6 months prior to baseline)
- Concomitant medications: record all medications have been taken at least once since one month prior to the baseline visit.
- Dose of Empagliflozin / DPP4-Inhibitor given
- PASS physician's electronic signature for data integrity

At visit 1, the patient will be requested to contact the treating physician in the event of any adverse events noted after initiating Empagliflozin or the comparator DPP-4 inhibitor treatment.

#### 9.2.2.2 Visit 2; 16±2 weeks from Visit 1

After 16±2 weeks from Visit 1, the patients will return for follow-up. The followings will be noted and recorded in the e-CRF.

- Visit date
- Physical examination: blood pressure, pulse rate, weight (if available)
- HbA1C (if available)
- Any change of Empagliflozin or comparator DPP-4 inhibitor given
- Concomitant anti-hyperglycemic agent including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)

- Concomitant medications including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Any adverse events noted
- Study completion status
- Discontinuation or continuation (if interruption, date of last administration, reason for interruption
- PASS physician's electronic signature for data integrity

#### 9.2.2.3 Visit 3; $32\pm2$ weeks from Visit 1

After 32±2 weeks from Visit 1, the patients will return for follow-up. The followings will be noted and recorded in the e-CRF.

- Visit date
- Physical examination: blood pressure, pulse rate, weight (if available)
- HbA1C (if available)
- Any change of Empagliflozin or comparator DPP-4 inhibitor given
- Concomitant anti-hyperglycaemic agent including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Concomitant medications including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Any adverse events noted
- Study completion status
- Discontinuation or continuation (if interruption, date of last administration, reason for interruption
- PASS physician's electronic signature for data integrity

#### 9.2.2.4 Visit 4; 52 weeks End of study

- Visit date
- Physical examination: blood pressure, pulse rate, weight
- HbA1C (if available)
- Any change of Empagliflozin or comparator DPP-4 inhibitor given
- Concomitant anti-hyperglycaemic agent including new medications taken since last visit: any change in the concomitant medications (dose and dosing intervals)
- Concomitant medications including new medications taken since last visit: any change in the concomitant medications ( dose and dosing intervals)
- Any adverse events noted
- Discontinuation or continuation (if interruption, date of last administration, reason for interruption

PASS physician's electronic signature for data integrity

#### 9.2.2.5 Follow-up period

Follow-up will start the day after the index date and last until end of study data (date of death or date of study end), the date during follow-up when specific exclusion criteria are met, the end date of the treatment of the index drug (Empagliflozin or other SGLT2 inhibitor or DPP-4 inhibitor) plus a defined grace period (30 days after the end of the last prescription's supply in main analyses), or the date on which a new treatment episode starts with any of the other index drugs.

Patients with adverse events noted at the final follow-up visit or upon premature discontinuation of Empagliflozin or the comparator DPP-4 inhibitor will be monitored further until the resolution of those adverse events. Alternatively, those patients will be followed up until the PASS physician and sponsor agree that no further follow-up is necessary.

#### 9.2.3 Study discontinuation

Boehringer Ingelheim reserves the right to discontinue the study overall or at a particular study site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular study site
- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the study, or any other administrative reasons.
- 3. Violation of Good Clinical Practice (GCP) (as applicable), the study protocol, or the contract by a study site or investigator, disturbing the appropriate conduct of the study

The investigator / the study site will be reimbursed for reasonable expenses incurred in case of study termination (except in case of the third reason).

#### 9.3 VARIABLES

#### **9.3.1** Safety

#### 9.3.1.1 Outcomes of safety

All reported adverse events in patients who take at least one dose of Empagliflozin or comparator DPP-4 inhibitor will be reported.

All documented information in the e-CRF will be analyzed at the end of the study. At the time of analysis, safety outcomes will be analyzed based on the current versions of MedDRA & BIcMQs

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.3.2 Exposures

The definition of drug exposure for Empagliflozin will be any patient using at least one prescription of Empagliflozin tablets (10 or 25 mg) or fixed-dose combinations with metformin. For the comparator group, the patients will have at least one prescription of DDP-4 inhibitors. DDP-4 inhibitor users included in this study will be using one of the following approved drugs in Saudi Arabia: Sitagliptin, Saxagliptin, Vildagliptin, Alogliptin, Linagliptin, or fixed-dose combinations of these drugs with metformin. [R17-3427] Furthermore, each member of the population exposed to Empagliflozin must have at least one prescription for Empagliflozin, with or without other glucose-lowering drugs (GLDs), and have no prior prescriptions of a DPP-4 inhibitor or Empagliflozin during the available preindex period. Each member of the population exposed to a DPP-4 inhibitor must have at least one prescription for a DPP-4 inhibitor, with or without other GLDs, and no prior prescriptions of a DPP-4 inhibitor or Empagliflozin during the available pre-index period. Add-on therapy will be allowed after using the exposure of interest as the initial drug for new users. Therefore, using the drug as part of dual therapy or triple therapy will be allowed. The use of studied medications will be defined on different levels: current use, recent use and discontinuation of the studied drugs. Current use of the index drugs will be defined from the date of prescription of Empagliflozin or DPP-4 inhibitor to the end of supply for that prescription plus a period of 30 days. Recent use will be defined from the end of current use (30 days after end of supply) until 90 days later (which is 120 days after end of supply). Discontinuation of the index drug will be defined as no further prescription 120 or more days after the end of the last prescription's supply. Patients who discontinue an index drug and then subsequently initiate another index drug will not be allowed to re-enter the study. Patients switching to or adding Empagliflozin to other antidiabetic medications will be compared to patients switching to or adding comparator treatment on the same background therapy. Identification of a "new-user" design is an appropriate method for studying secondline therapies in chronic conditions.

During the statistical analyses, analyses will be stratified by treatment complexity (mono vs. dual vs. triple therapy) and by calendar time of treatment initiation. Prior or current use of insulin is allowed; an additional stratified analysis by insulin use is planned. Propensity scores based on information prior to the index date will be used to account for potential confounding.

#### 9.3.3 Outcomes

This study proposed to assess and evaluate the risk of ketoacidosis, severe urinary tract infections, volume depletion and dehydration associated with the use of Empagliflozin compared with the use of DPP-4 inhibitors in T2DM. As per ADA, ketoacidosis is defined as a serious condition because of inability of body cells to get glucose as a source of energy, and subsequently, the body produces ketones as the result of burning fat for energy. DKA occurs because of a lack of insulin in the body, not enough food intakes in diabetic patients and insulin reaction (low blood glucose). It is characterized by high ketones levels, positive ketones in the urine and high pH levels. Specifically, for the SGLT2i induced DKA the blood glucose level may not be increased above 240 mg/dl. [R17-3411] ¬The second outcome, which is severe urinary tract infection, is defined as pyelonephritis or urosepsis. Volume

depletion is the reduction in the extracellular fluids. This differs from dehydration, which is the loss of total body water that leads to hypertonicity. To ascertain the outcome diagnosis, signs and symptoms along with the laboratory tests results will be used.

All identified primary outcomes will be evaluated also during the period of the month of Ramadan.

#### 9.3.4 Covariates

The covariates of interest are age, gender, body mass index (BMI), blood pressure, blood glucose level, and HbA1c, if available. Comorbidities of interest include hypertension, dyslipidaemia, kidney diseases, kidney stones, history of kidney transplant, liver diseases, prostate diseases, pancreatitis, surgery, infections (other than UTIs) and heart diseases, if available. In addition, genital defects, urinary tract anatomical defects, lab variables (CBC, FPG, OGTT, ketones level, amylase, lipase, arterial blood gas, pH, bicarbonate, ScCr, lipid profile tests, BUN, liver tests, INR and platelets) and concomitant medications

will be considered as covariates. All these covariates will be identified, if available, for all cohort members prior to and including the index date. Severity of T2DM will be assessed by HbA1c values, concomitant diagnoses and duration since the first diagnosis, when available.

These and other variables that can differ by exposure group will be considered for inclusion as predictors in the logistic regression models used to generate the propensity scores. Propensity scores will be used in the analysis to quantify the probability of receiving Empagliflozin at the index date for new users of both Empagliflozin and DPP-4 inhibitors. At the index date, cohort members will also be classified by indicator variables on the calendar time of cohort entry (by quarter) whether the index treatment (Empagliflozin or DPP-4 inhibitor) was added to existing medication (adding on), or if the index treatment was initiated as a replacement for another GLD (switching from the existing GLD to Empagliflozin or DPP-4 inhibitor), and whether this treatment was received as monotherapy or as dual or triple therapy. A variable indicating whether or not patients were receiving insulin at the index date will also be created.

List of Variables, (other variables will be added during the study period) Demographics

- 1. Age
- 2. Gender

Hospitalization, when available

- 3. Admission date
- 4. Place admitted from
- 5. Outcomes diagnosis date
- 6. Place of diagnosis (ER, Inpatients, Outpatient)

#### Treatment

- 7. Treatment initiation date
- 8. Treatment discontinuation date

#### Outcomes, when available

- 9. Date of DKA diagnosis
- 10. Date of UTI diagnosis
- 11. Date of dehydration diagnosis
- 12. Date of volume depletion diagnosis
- 13. Date of death
- 14. Primary cause of death
- 15. Date of discharge
- 16. Date of admission
- 17. Reason for admission

#### Lab variables / Vital signs, when available

- 18. Weight
- 19. Height
- 20. CBC
- 21. Blood glucose
- 22. HbA1c
- 23. FPG
- 24. OGTT
- 25. Ketones (Urine and/or blood)
- 26. Blood pressure
- 27. Amylase
- 28. Lipase
- 29. Triglyceride (TG)
- 30. Liver function tests
- 31. Arterial blood gas
- 32. pH
- 33. Bicarbonate
- 34. Lipid profile tests
- 35. INR
- 36. eGFR
- 37. CrCl
- 38. ScCr
- 39. BUN

#### Comorbidities, Medical History

- 40. Diabetes
- 41. Kidney diseases
- 42. Hypertension
- 43. Heart failure
- 44. Acute coronary diseases
- 45. Heart diseases
- 46. Diabetic ketoacidosis

- 47. Pregnancy
- 48. Abdominal trauma
- 49. Kidney stones
- 50. Body paralysis (paraplegia or quadriplegia)
- 51. Pancreatitis
- 52. Dyslipidaemia
- 53. Cerebrovascular disease
- 54. Pulmonary disease
- 55. Hypothyroidism
- 56. Hyperthyroidism
- 57. Surgery
- 58. Liver disease
- 59. HIV/AIDS
- 60. Cancer
- 61. Hepatitis "A,B,C"
- 62. Cholestatic hepatitis
- 63. Acute liver disease
- 64. Liver cirrhosis
- 65. Kidney transplant
- 66. Prostate diseases
- 67. Burns
- 68. Genital defects
- 69. Urinary tract anatomical defects
- 70. Other liver diseases

Prior medications exposure in the last 6 months and during the study period

- 71. Empagliflozin
- 72. Sitagliptin
- 73. Saxagliptin
- 74. Vildagliptin
- 75. Alogliptin
- 76. Linagliptin
- 77. Insulin (all types)
- 78. Metformin (single or combination)
- 79. Sulfonylureas
- 80. Meglitinides
- 81. Thiazolidinediones
- 82. α-glucosidase inhibitors
- 83. Glucagon-like peptide-1 receptor agonist
- 84. Lipid lowering agents (Statins, Fibrates, Niacin)
- 85. Antihypertensive agents (Diuretics, ACEIs, B-blocker)
- 86. Antipsychotic medications
- 87. Corticosteroids

#### 9.4 DATA SOURCES

This study will be carried out in the manner of successive survey that the investigator will be asked to successively write in the case report forms (e-CRFs) from the subject who was initially administered the drug following the study start date to the requested number of subjects without omission. Prior to initiation of the study, a written contract shall be concluded, with the head of the site or the investigator with his/her consent for non-interventional study with new data collection.

This study will be carried out in the manner of successive surveys where the investigator will be asked to write in the case report forms (e -CRFs). Number of recruited patients will be comparable in each group within a given timeframe (i.e each site will ensure to recruit similar number of patients for each group according to assigned blocks of enrolment). Data on the period preceding the index date will be collected at the time of the first survey.

The site(s) will be primary care clinics, hospital clinics and other outpatient clinics. Data from hospitals will be documented when needed, especially if there are cases of admission for one of the study outcomes. Discharge data will always be documented by the investigator when needed.

Demographics (age, gender), comorbidities (cardiac, hepatic, oncologic, renal, neurologic, immunologic, respiratory and vascular), previous and current hypoglycaemic agent exposures (biguanides, sulfonylureas, meglitinides, thiazolidinediones, dipeptidyl peptidase-4 inhibitors, α-glucosidase inhibitors, glucagon-like peptide-1 receptor agonists and insulin), and laboratory data (complete blood count, blood glucose level "all available types", and HbA1c) variables will be obtained from either the medical record or during the first survey (Section 9.3.4).

#### 9.5 STUDY SIZE

The sample size is of 1500 patients; it is based on SFDA requirements. As per SFDA regulation and requirements to detect the DKA cases, 750 patients will be enrolled in each group (DPP4i and SGLT-2i). The number of recruited patients will be comparable in each group within a given time frame (i.e. each site will ensure to recruit similar number of patients for each group according to assigned blocks of enrolment). In addition, prevalence of the primary outcomes was searched in literature and a study found assuming the prevalence to be around 25% (urinary tract infection and other risk factors) among Saudi patients with diabetes.

#### 9.6 DATA MANAGEMENT

Patients' data will be gathered by e-CRF. The data management procedures to ensure the quality of the data are described in detail in the data management plan (DMP) available in TMF. Data management and statistics will be outsourced to a qualified contract research organization (CRO).

#### 9.7 **DATA ANALYSIS**

Details of all analyses and variables specification will be defined in a separate SEAP.

Patients are grouped according the exposure to either Empagliflozin or DPP-4 inhibitors. Data will be analysed per group. Let the index period define the time from index date to the end of treatment as defined in section 9.3.2 by current use, and the follow-up period the time from index date to the end of observation as defined in section 9. Incidences will be derived if events of interest occur in the respective period. The main analysis will consider index periods only, a secondary analysis will consider only the time of the index period in the month of Ramadan in every year, while sensitivity analyses will consider respective follow-up periods, overall or during Ramadan only. Times from index date to first occurrence will also be determined per event of interest and described by means of Kaplan-Meier estimates and median times with 95% confidence intervals, where appropriate.

All individual data will be listed and described per group by means of summary tables presenting frequency counts and percentages for categorical data and arithmetic means, standard deviations, medians, minimum and maximum values for continuous data. Baseline is defined as the last observation on or before the index date.

For the assessment of the primary and secondary objectives, the main data analysis will be conducted in two stages:

- 1) Construction of the PS by modelling the exposure to Empagliflozin vs. DPP-4 inhibitor;
- 2) Estimation of the effect of exposure to Empagliflozin on the risk of ketoacidosis, severe urinary tract infections, volume depletion and dehydration compared to those exposed to DPP-4 inhibitor.

Propensity score stratification will be the primary method to control for the confounders in the analysis phase. The stratification will divide the study population in several groups (max. 5 groups) based on their propensity score value. Propensity score matching will also be used as secondary method in the analysis phase.

All statistical tests will be conducted with a two-sided significance level alpha of 0.05 and all analyses will be conducted using SAS statistical analysis software version 9.4 (SAS Institute, Inc., Cary, NC) or later.

#### 9.7.1 Propensity score modelling

A propensity score (PS) method will be utilized to control for confounding in the analysis phase. It is used to balance the baseline covariates predictive of treatment, to lessen the unequal chance of receiving Empagliflozin versus DDP-4 inhibitors. PS will be estimated with logistic regression for each cohort member. PS is one of effective methods used in epidemiological studies analyses.

Bivariate analysis will be initially used for the selection of potential clinical covariates for inclusion in the propensity score model. Demographic and clinical categorical data will be analysed using an  $\chi^2$  or Fisher's exact test while continuous variables will be analysed using a student's t-test or Mann-Whitney U test.

The model will be selected in a process optimizing the goodness of fit. Only clinically relevant, statistically significant (p-value <0.25) covariates will be included. Propensity

scores will be stratified into quintiles, and subsequent covariate balance will be reviewed graphically and with Mantel-Haenszel tests.

#### 9.7.2 Main analysis using stratification

For the incident users of Empagliflozin along with their respective comparators, analysis will be performed using the "as-treated" (AT) approach. This corresponds to censoring individuals who discontinue use of the index drug, i.e. who either switch from the index drug to any other of the index drugs (Empagliflozin or DPP-4 inhibitor) during follow-up or who stop using the index drug. The AT approach is considering index periods. For each event of interest, ketoacidosis, severe urinary tract infections, volume depletion, and dehydration, crude and adjusted incidence rates per cohort will be described and compared by means of incidence rate ratios (IRR). Incidence rates will be reported as point estimates and 95% confidence intervals (CIs). Crude incidence rates will be adjusted per 1,000 personyears. Per cohort and, where appropriate per stratum and/or subgroup, the number of personyears is the sum of length of index periods of all patients. Time to first event occurrence will be compared by means of hazard ratios and their 95% confidence intervals.

IRRs and hazard ratios are analysed using stratification. Strata are defined by PS quintiles. IRRs are investigated by means of a stratified Mantel-Haenszel analysis, while hazard ratios are investigated by means of a Cox regression, if proportional hazards can be assumed.



#### 9.8 QUALITY CONTROL

All entries in the e-CRF and the existing coding will be stored in a database. The structure of the database is based on the division into sections and entry fields defined in the e-CRF. To improve and ensure data quality, data checks will be performed automatically in the e-CRF directly on electronic entry at the study site.

Plausible value ranges for numerical data entries and logical data and list entries will be filed in the e-CRF. The tests for consistency and completeness based on this will be performed during entry in the e-CRF. The validity of the recorded data will therefore be ensured by the validations incorporated in the documentation system, which highlight incorrect or implausible entries to the data entry clerk/doctor.

If corrections are necessary after the data are saved, these will be documented in an audit trail.

For the further quality assurance of the documented patient observations, a sample-based source data comparison will be performed on about 10% of the sites. An additional inspection/quality assurance check of this PASS can be performed in case of any deviation.

#### 9.9 LIMITATIONS OF THE RESEARCH METHODS

There are several methodological challenges when conducting epidemiologic studies to evaluate the association between glucose-lowering medications and outcomes of interest among patients with diabetes. These challenges include, but are not limited to, changes in treatment in response to advancing diabetes or due to adverse effects of specific drugs and time-varying risk of an outcome depending on duration of exposure

Another limitation is that, the number of patients may be low to assess the risk of DKA.

Some patients may discontinue the study before Ramadan period and will not contribute to the assessment of the safety during this period.

#### 9.10 OTHER ASPECTS

#### 9.10.1 Data quality assurance

A quality assurance audit/inspection of this study may be conducted by the sponsor or sponsor's designees or by Institutional Review Board (IRBs) / Independent Ethics Committee (IECs) or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's study-related files and correspondence, and the informed consent documentation of this study.

#### 9.10.2 Study records

Case Report Forms (e-CRFs) for individual patients will be provided by the sponsor, either on paper or via remote data capture.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 9.10.2.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data reported on the e-CRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the study; also current medical records must be available.

For paper e-CRFs, the following data need to be derived from source documents:

- Patient identification (gender, date of birth)
- Patient participation in the study (substance, study number, patient number, date patient was informed)
- Dates of Patient's visits, including prescription of study medication
- Medical history (including study indication and concomitant diseases, if applicable)
- Medication history
- Adverse events and outcome events (onset date (mandatory), and end date (if available))
- Serious adverse events (SAEs) (onset date (mandatory), and end date (if available))
- Concomitant therapy (start date, changes)
- Originals or copies of laboratory results (in validated electronic format, if available)
- Conclusion of Patient's Participation in the study

#### 9.10.2.2 Direct access to source data and documents

The investigator / institution will permit study-related monitoring, audits, IRB / IEC review and regulatory inspection, providing direct access to all related source data / documents. e-CRFs and all source documents, including progress notes and copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical study monitor, auditor and inspection by health authorities (e.g. US Food and Drug Administration (FDA)). The Clinical Research Associate (CRA) / Clinical Monitor Local (CML) and auditor may review all e-CRFs and written informed consents. The accuracy of the data will be verified by reviewing the documents described in Section 9.10.2.1.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 10. PROTECTION OF HUMAN SUBJECTS

The study will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki, in accordance with the ICH Harmonized Tripartite Guideline for Good Clinical Practice (GCP) (to the extent applicable to the NIS setting and required by local regulations), Good Epidemiological Practice (GEP), Guidelines for Good Pharmacoepidemiology Practice (GPP), and relevant BI and/or CRO Standard Operating Procedures (SOPs). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study subjects against any immediate hazard, and also of any serious breaches of the protocol/ICH GCP.

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

The protocol of this regulatory requisite PASS will be submitted to Saudi FDA for review and approval. This study will be conducted in accordance with the SFDA guidelines of good pharmacovigilance practice version 2.0.

will submit periodic reports as per SFDA guidelines of good pharmacovigilance practice version 2.0, and the final report to SFDA upon study completion. The periodic report for the final year will be substituted with the final report.

## 10.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This study will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and Competent Authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the study, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the investigator as part of the study records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

The patient must be informed that his/her personal study-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorised monitors (CML/CRA) or Quality Medicine auditors appointed by Boehringer Ingelheim, by appropriate IRB / IEC members, and by inspectors from regulatory authorities.

#### 10.2 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this study is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the study need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities <for EU>, *i.e.* the CA.

# 11. MANAGEMENT AND REPORTING OF ADVERSE EVENTS/ADVERSE REACTIONS

#### 11.1 DEFINITION OF ADVERSE EVENTS

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence in a patient or clinical investigation subject administered a medicinal product and which does not necessarily have a causal relationship with this treatment. An adverse event can therefore be any unfavorable and unintended sign (e.g. an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### Adverse reaction

An adverse reaction is defined as a response to a medicinal product which is noxious and unintended. Response in this context means that a causal relationship between a medicinal product and an adverse event is at least a reasonable possibility. Adverse reactions may arise from use of the product within or outside the terms of the marketing authorization or from occupational exposure. Conditions of use outside the marketing authorization include off-label use, overdose, misuse, abuse and medication errors.

#### Serious adverse event

A serious adverse event is defined as any AE which

- results in death,
- is life-threatening,
- requires in-patient hospitalization, or
- prolongation of existing hospitalization,
- results in persistent or significant disability or incapacity, or
- is a congenital anomaly/birth defect

Life-threatening in this context refers to a reaction in which the patient was at risk of death at the time of the reaction; it does not refer to a reaction that hypothetically might have caused death if more severe.

Medical and scientific judgment should be exercised in deciding whether other situations should be considered serious reactions, such as important medical events that might not be immediately life threatening or result in death or hospitalisation but might jeopardize the patient or might require intervention to prevent one of the other outcomes listed above.

Examples of such events are intensive treatment in an emergency room or at home for allergic bronchospasm, blood dyscrasias or convulsions that do not result in hospitalisation or development of dependency or abuse. Any suspected transmission via a medicinal product of an infectious agent is also considered a serious adverse reaction.

Table 1: Clinical criteria for Adverse Event of Special Interest

| Endpoint | Definition |
|---|---|
| Acute liver injury | Any the following criteria: An elevation of AST and/or ALT $\geq$ 3-fold ULN combined with an elevation of bilirubin $\geq$ 2-fold ULN measured in the same blood draw sample. An isolated elevation of AST and /or ALT $\geq$ 5-fold ULN irrespective of any bilirubin elevation |
| Decreased renal function | Creatinine value shows $a \ge 2$ -fold increase from baseline and is above the upper limit of normal (ULN) |
| ketoacidosis and diabetic<br>ketoacidosis (DKA) | Defined as a serious condition because of inability of body cells to get glucose as a source of energy, and subsequently, the body produces ketones as the result of burning fat for energy. DKA occurs because of a lack of insulin in the body, not enough food intakes in diabetic patients and insulin reaction (low blood glucose). It is characterized by high ketones levels, positive ketones in the urine and high pH levels. Specifically, for the SGLT2i induced DKA the blood glucose level may not be increased above 240 mg/dl. |
| Events involving lower<br>limb amputation | This definition includes amputation (i.e. resection of a limb through a bone), disarticulation (i.e. resection of a limb through a joint) and auto-amputations (i.e. spontaneous separation of non-viable portion of the lower limb). Not included in this definition are debridement (removal of callus or dead tissue), procedures on a stump (like stump revision, drainage of an abscess, wound revision etc.) and other procedures (e.g., nail resection or removal) without a concomitant resection of a limb (amputation or disarticulation)." Request to report each lower limb amputation as separate AE |

ALT = alanine aminotransferase; ULN = upper limit of normal range.

## 11.2 ADVERSE EVENT AND SERIOUS ADVERSE EVENT COLLECTION AND REPORTING

The investigator shall maintain and keep detailed records of all AEs in their patient files.

#### Collection of AEs

The study design is of non-interventional nature and the study is conducted within the conditions of the approved marketing authorization.

The following must be collected by the investigator in the e-CRF from signing the informed consent onwards until the end of the study:

All adverse events

All AEs, including those persisting after study completion must be followed up until they are resolved, have been sufficiently characterized, or no further information can be obtained.

The investigator carefully assesses whether an AE constitutes an ADR using the information below.

AEs considered "Always Serious"

In accordance with the European Medicines Agency initiative on Important Medical Events, BI has set up a list of AEs, which by their nature, can always be considered to be "serious" even though they may not have met the criteria of an SAE as given above.

The latest list of "Always Serious AEs" can be found in the ISF. These events should always be reported in the eCRF as SAEs as described above.

Note: Cancers of new histology and exacerbations of existing cancer must be reported as a serious event regardless of the duration between discontinuation of the drug and the occurrence of the cancer.

#### Causal relationship of adverse event

The definition of an adverse reaction implies at least a reasonable possibility of a causal relationship between a suspected medicinal product and an adverse event. An adverse reaction, in contrast to an adverse event, is characterized by the fact that a causal relationship between a medicinal product and an occurrence is suspected.

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history.

Arguments that may suggest a reasonable causal relationship could be:

- The event is **consistent with the known pharmacology** of the drug
- The event is known to be caused by or attributed to the drug class.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

- A plausible time to onset of the event relative to the time of drug exposure.
- Evidence that the **event is reproducible** when the drug is re-introduced
- **No medically sound alternative etiologies** that could explain the event (e.g. preexisting or concomitant diseases, or co-medications).
- The event is typically **drug-related and infrequent in the general population** not exposed to drugs (e.g. Stevens-Johnson syndrome).
- An indication of dose-response (i.e. greater effect size if the dose is increased, smaller effect size if dose is diminished).

Arguments that may suggest that there is **no reasonable possibility of a causal relationship** could be:

- No plausible time to onset of the event relative to the time of drug exposure is evident (e.g. pre-treatment cases, diagnosis of cancer or chronic disease within days/weeks of drug administration; an allergic reaction weeks after discontinuation of the drug concerned)
- Continuation of the event despite the withdrawal of the medication, taking into
  account the pharmacological properties of the compound (e.g. after 5 half-lives).
   Of note, this criterion may not be applicable to events whose time course is prolonged
  despite removing the original trigger.
- Additional arguments amongst those stated before, like alternative explanation (e.g. situations where other drugs or underlying diseases appear to provide a more likely explanation for the observed event than the drug concerned).
- Disappearance of the event even though the study drug treatment continues or remains unchanged.

#### Intensity of adverse event

The intensity of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated Moderate: Enough discomfort to cause interference with usual activity

Severe: Incapacitating or causing inability to work or to perform usual activities

#### Pregnancy:

In rare cases, pregnancy might occur in a study. Once a subject has been enrolled into the study, after having taken Jardiance, the investigator must report any drug exposure during pregnancy, which occurred in a female subject or in a partner to a male subject to the Sponsor by means of Part A of the Pregnancy Monitoring Form. The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up and reported by means of Part B of the Pregnancy Monitoring Form.

In the absence of a reportable AE, only the Pregnancy Monitoring Form must be completed, otherwise the NIS AE form is to be completed and forwarded as well within the respective timelines.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

Table 2: Expedited Reporting of AEs and Drug Exposure During Pregnancy

The following must be reported by the investigator on the NIS AE form from signing the informed consent onwards until the end of the study:

| Type of Report | Timeline |
|---|---|
| All Serious Related Adverse Events (SAEs) with Jardiance®, Trajenta® and/or Synjardy® | immediately within 24 hours |
| Adverse Event of Special interest associated with Jardiance® | immediately within 24 hours |
| All AEs with fatal outcome in patients exposed to Jardiance®, Trajenta® and/or Synjardy® | immediately within 24 hours |
| All non-serious Related Adverse Events associated with Jardiance®, Trajenta® and/or Synjardy® | 7 calendar days |
| All pregnancy associated with Jardiance®, Trajenta® and/or Synjardy® on pregnancy monitoring forms | 7 calendar days |

The same timelines apply if follow-up information becomes available for the respective events. In specific occasions the Investigator could inform the Sponsor upfront via telephone. This does not replace the requirement to complete and secure email or fax the NIS AE form.

#### Reporting of DKA cases:

An additional information will be requested with a targeted form.

#### Information required

For each reportable adverse event, the investigator should provide the information requested on the appropriate e-CRF pages and the NIS AE form.

#### Reporting of related Adverse Events associated with any other BI drug

The investigator is encouraged to report all adverse events related to any BI drug other than **Jardiance®**, **Trajenta®** and/or **Synjardy®** according to the local regulatory requirements for spontaneous AE reporting at the investigator's discretion by using the locally established routes and AE report forms. The term AE includes drug exposure during pregnancy, and, regardless of whether an AE occurred or not, any abuse, off-label use, misuse, medication error, occupational exposure, lack of effect, and unexpected benefit.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

#### 11.3 REPORTING TO HEALTH AUTHORITIES

Adverse event reporting to regulatory agencies will be done by the MAH according to local and international regulatory requirements.

Proprietary confidential information © 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies

# 12. PLANS FOR DISSEMINATING AND COMMUNICATING STUDY RESULTS

The rights of the investigator and of the sponsor with regard to publication of the results of this study are described in the investigator contract. As a general rule, no study results should be published prior to finalization of the Study Report.

#### 13. REFERENCES

#### 13.1 PUBLISHED REFERENCES

| P17-11212 | Blair M. Diabetes Mellitus Review. Urol Nurs. 2016;36(1):27-36. |
|---|---|
| R16-4703 | The International Diabetes Federation (IDF). Diabetes Atlas. Seventh Edition. 2015. http://www.diabetesatlas.org/ Accessed on July-2016. |
| R17-3422 | Statistics about Diabetes. American Diabetes Association. http://www.diabetes.org/diabetes-basics/statistics/. Accessed on July-2016. |
| P14-06594 | Liakos A, Karagiannis T, Athanasiadou E, et al. Efficacy and safety of Empagliflozin for type 2 diabetes: a systematic review and meta-analysis. Diabetes Obes Metab. 2014;16(10):984-93. |
| P16-06686 | Monica Reddy RP, Inzucchi SE. SGLT2 inhibitors in the management of type 2 diabetes. Endocrine. 2016;53(2):364-72. |
| R17-3413 | Empagliflozin. Summary Product Characteristics. Electronic Medicines Compendium. https://www.medicines.org.uk/emc/medicine/28973. Accessed on July-2016. |
| P15-03461 | Kadowaki T, Haneda M, Inagaki N, et al. Efficacy and safety of Empagliflozin monotherapy for 52 weeks in Japanese patients with type 2 diabetes: a randomized, double-blind, parallel-group study. Adv Ther. 2015;32(4):306-18. |
| P13-09179 | Kovacs CS, Seshiah V, Swallow R, et al. Empagliflozin improves glycaemic and weight control as add-on therapy to pioglitazone or pioglitazone plus metformin in patients with type 2 diabetes: a 24-week, randomized, placebocontrolled trial. Diabetes Obes Metab. 2014;16(2):147-58. |
| P15-05613 | Merker L, Haring HU, Christiansen AV, et al. Empagliflozin as add-on to metformin in people with Type 2 diabetes. Diabet Med. 2015;32(12):1555-67. |
| R17-3412 | Empagliflozin. Drug Databases. Food and Drug Administration. http://www.accessdata.fda.gov/drugsatfda_docs/label/2016/204629s005lbl.pdf Accessed on July-2016. |

P15-01744 Dailey G. Empagliflozin for the treatment of type 2 diabetes mellitus: An overview of safety and efficacy based on Phase 3 trials. J Diabetes. 2015;7(4):448-61.

P15-09840 Zinman B, Wanner C, Lachin JM, et al. Empagliflozin, Cardiovascular Outcomes, and Mortality in Type 2 Diabetes. N Engl J Med. 2015;373(22):2117-28.

P16-01253 Fitchett D, Zinman B, Wanner C, et al. Heart failure outcomes with Empagliflozin in patients with type 2 diabetes at high cardiovascular risk: results of the EMPA-REG OUTCOME® trial. Eur Heart J. 2016;37(19):1526-34.

R17-3410 ADA. American Diabetes Association. Standards of medical care in diabetes—2016. Diabetes Care. 2016;39(suppl 1):S1-S106. http://care.diabetesjournals.org/content/39/Supplement\_1 . Accessed on August/2016.

P13-09179 ICD-9-CM Diagnosis Codes. Endocrine, nutritional and metabolic diseases. Icd9data. http://www.icd9data.com/2014/Volume1/240-279/249-259/250/. Accessed on August/2016.

R17-3428 ICD-10-CM Diagnosis Codes. Endocrine, nutritional and metabolic diseases. Icd10data. http://www.icd10data.com/ICD10CM/Codes/E00-E89/E08-E13/E11-. Accessed on August/2016.

R17-3427 Saudi Drug List. Saudi Food and Drug Authority. http://www.sfda.gov.sa/en/drug/search/Pages/default.aspx . Accessed on August/2016.

R17-3411 DKA (Ketoacidosis) & Ketones. American Diabetes Association. http://www.diabetes.org/living-with-diabetes/complications/ketoacidosis-dka.html?referrer=https://www.google.com.sa/

